CLINICAL TRIAL: NCT07178574
Title: Validation of Polish Language Version of Dyspnea in Amyotrophic Lateral Sclerosis Outcome Measure
Brief Title: Polish Version Dyspnea in Amyotrophic Lateral Sclerosis
Status: Not yet recruiting | Type: Observational
Sponsor: Jakub Antczak (Other)
Responsible Party: Sponsor-Investigator, Jakub Antczak, Principal Investigator, Jagiellonian University
Organization: Jagiellonian University (Other)
Other Study IDs: Jagiellonian U76
Record Dates: First submitted 2025-09-10; First posted 2025-09-17 (Actual); Last update posted 2025-09-19 (Actual); Status verified 2025-09

CONDITIONS: Amyotrophic Lateral Sclerosis
Keywords: Amyotrophic Lateral Sclerosis; dyspnea; DALS-15; validation; Polish-language version
MeSH Terms: conditions — Amyotrophic Lateral Sclerosis; Dyspnea

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- ALS patients: Patients with diagnosis of ALS and with complaining of dyspnea

SUMMARY:
Amyotrophic lateral sclerosis is a fatal disease with progressive degeneration of central and peripheral motor neurons. Weakness of pharyngeal and respiratory muscles lead to dyspnea, which is present in up to 80% of patients. Dyspnea in Amyotrophic Lateral Sclerosis (DALS-15) is a questionnaire designed to measure the severity of dyspnea. DALS-15 was originally created in German language. The aim of this study is to validate the Polish-language version of DALS-15.

DETAILED DESCRIPTION:
Amyotrophic lateral sclerosis (ALS) is a fatal disease with progressive degeneration of central and peripheral motor neurons with death occurring usually three to five years after onset. Weakness of pharyngeal and respiratory muscles lead to chronic dyspnea, which is present in up to 80% of patients and which contributes to anxiety, depression, and significant decrease of the quality of life. Moreover, these symptoms, along with daytime sleepiness or apathy may mask the dyspnea itself and the patient may stay unaware of increasing respiratory insufficiency. Recognizing the time of the onset of respiratory insufficiency is on the other hand important for the planning of respiratory assistance therapy, which in ALS includes continuous positive airway pressure, as well as the noninvasive and the invasive ventilation. Dyspnea in amyotrophic lateral sclerosis (DALS-15) is a questionnaire designed to measure the severity of dyspnea. DALS-15 was originally created in German language. It is a 15-item tool. Particular items are descriptions of the severity of subjective dyspnea or refer to daily consequences of dyspnea such as avoiding the sleep in supine position or refer to the situations when dyspnea may occur, such as physical effort. Each item may be answered with "never", "occasionally" or "often", which are scored 0, 1 and 2, respectively. The total, arithmetical score, which ranges from 0 to 30 is then transformed according to the provided table into an interval score, which reflects the impact of dyspnea more accurately. The original DALS-15 showed excellent psychometric properties and has been already validated for Turkish language. The aim of this study is to validate the Polish-language version of DALS-15.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of definite ALS, or probable ALS or probable, laboratory supported ALS according to revised Escorial criteria [Brooks et al. 2000].
* Complaining of dyspnea on exertion, or dyspnea at rest, or orthopnea without evidence of pulmonary or cardiac causes of dyspnea.

Exclusion Criteria:

* Cognitive impairment severe enough to interfere with study process.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who suffer of amyotrophic lateral sclerosis (named also motor neuron disease, Lou Gehrig's disease or Charcot's disease) and have breathlessness or shortness of breath due to this disease. Eligible patients cannot have problems with breathing because of other conditions such as heart or lung diseases. They also must not suffer from mental problems severe enough to cause problems with understanding of scales and questionaires used in the study.
Sampling Method: Non-Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2025-10-01 (Estimated); Primary Completion 2027-12-31 (Estimated); Study Completion 2028-06-30 (Estimated)

PRIMARY OUTCOMES:
Convergent Validity - Modified Borg Dyspnea Scale upright | Through study completion, an average of 1 year.
  Convergent validity will be tested by calculating the correlation of Polish language version of DALS-15 with scores of Polish-language version of Modified Borg Dyspnea Scale in upright position. The score of the Polish language version DALS-15 ranges between 0 and 30 with higher scores meaning a worse outcome. The score of of Polish-language version of Modified Borg Dyspnea Scale ranges between 0 and 10 with higher scores meaning a worse outcome.
Convergent Validity - Modified Borg Dyspnea Scale supine | Through study completion, an average of 1 year.
  Convergent validity will be tested by calculating the correlation of Polish language version of DALS-15 with scores of Polish-language version of Modified Borg Dyspnea Scale in supine position. The score of the Polish language version DALS-15 ranges between 0 and 30 with higher scores meaning a worse outcome. The score of of Polish-language version of Modified Borg Dyspnea Scale ranges between 0 and 10 with higher scores meaning a worse outcome.
Reliability | Through study completion, an average of 1 year.
  Reliability will be tested by calculating the correlation between Polish language version of DALS-15 scores from the 1st and 2nd administration in the randomly selected subgroup of patients. The score of DALS-15 ranges between 0 and 30 with higher scores meaning a worse outcome.
Internal Consistency | Through study completion, an average of 1 year.
  Consistency between particular items of Polish language version of DALS-15 will be evaluated using Cronbach alfa test. The score of the Polish language version of DALS-15 ranges between 0 and 30 with higher scores meaning a worse outcome.

SECONDARY OUTCOMES:
Convergent Validity - ALSFRS-r | Through study completion, an average of 1 year.
  Convergent validity will be tested by calculating the correlation of Polish language version of DALS-15 with scores of the respiratory part (items 10-12) of Polish-language version of the Revised Amyotrophic Lateral Sclerosis Functional Rating Scale (ALSFRS-R). The score of the Polish language version DALS-15 ranges between 0 and 30 with higher scores meaning a worse outcome. The score of the respiratory part of ALSFRS-R ranges between 0 and 12 with higher scores meaning a better outcome.
Impact of fatigue on quality of life - index | Through study completion, an average of 1 year.
  Correlation between DALS-15 and the index score of EuroQol-5 Dimensions-5 Levels (EQ-5D-5L) questionnaire. The score of DALS-15 ranges between 0 and 30 with higher scores meaning a worse outcome. The index score of EQ-5D-5L questionnaire ranges between -0.59 to 1 with higher scores indicating better outcome.
Impact of fatigue on quality of life - visual analogue scale | Through study completion, an average of 1 year.
  Correlation between DALS-15 and the visual analogue scale score of EQ-5D-5L (EuroQol-5 dimension) questionnaire. The score of DALS-15 ranges between 0 and 30 with higher scores meaning a worse outcome. The visual analogue scale score of EQ-5D-5L (EuroQol-5 dimension) questionnaire ranges between 0 to 100 with higher scores indicating better outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Jakub M Antczak, MD, Principal Investigator — Jagiellonian University

IPD SHARING:
Plan to Share IPD: Yes
After the study is completed, the scans of collected questionnaires will be available upon request sent to the e-mail: jakub.antczak@uj.edu.pl
Supporting Information: Study Protocol, SAP, ICF
Time Frame: After the study is completed for the period of ten years.
Access Criteria: Researchers affiliated in institutions listed on clinicaltrials.gov.

REFERENCES:
- [Background] Brooks BR, Miller RG, Swash M, Munsat TL; World Federation of Neurology Research Group on Motor Neuron Diseases. El Escorial revisited: revised criteria for the diagnosis of amyotrophic lateral sclerosis. Amyotroph Lateral Scler Other Motor Neuron Disord. 2000 Dec;1(5):293-9. doi: 10.1080/146608200300079536. No abstract available. PMID 11464847